CLINICAL TRIAL: NCT01212744
Title: A Phase 2, Open-Label Study to Evaluate the Safety, Tolerability, and Efficacy of Subcutaneous Dose Levels of rAvPAL-PEG Administered Daily in Subjects With Phenylketonuria
Brief Title: Safety, Tolerability, and Efficacy Study of rAvPAL-PEG Administered Daily in Subjects With Phenylketonuria (PKU)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAL-004
Record Dates: First submitted 2010-09-29; First posted 2010-10-01 (Estimated); Results first posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Phenylketonuria
Keywords: PEG PAL; PKU; injection;
MeSH Terms: conditions — Phenylketonurias | interventions — pegvaliase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rAvPAL-PEG (Experimental): rAvPAL-PEG in varying doses
  Interventions: Drug: rAvPAL-PEG

INTERVENTIONS:
Drug: rAvPAL-PEG — 0.06 mg/kg/day, 0.1 mg/kg/day, 0.2 mg/kg/day, 0.4 mg/kg/day, 0.6 mg/kg/day, 0.8 mg/kg/day
  Other Names: Recombinant Anabaena variabilis phenylalanine ammonia lyase

SUMMARY:
The purpose of this study is to evaluate the effect of daily administration of rAvPAL-PEG on the reduction of blood Phe concentrations in subjects with PKU.

DETAILED DESCRIPTION:
This 16-week multi-center, open-label, Phase 2 study is designed to evaluate the safety, tolerability,and efficacy of daily SC injections of rAvPAL-PEG in subjects with PKU. Subjects who are naïve to prior treatment with rAvPAL-PEG and who have met the other study eligibility criteria will be enrolled at approximately 8 sites in the US and Canada. Up to 6 daily dose levels of rAvPAL-PEG are planned and may be assessed during this study (0.06 mg/kg/day, 0.1 mg/kg/day, 0.2 mg/kg/day;0.4 mg/kg/day, 0.6 mg/kg/day, or 0.8 mg/kg/day). Enrollment will begin with the 0.4 mg/kg/day dose level and additional higher or lower doses may be added. The additional dose levels chosen for assessment will be based on the safety (systemic reaction or clinically significant abnormal laboratory test results assessed as related to study drug) and efficacy (blood Phe reduction to less than or equal to 60 μmol/L) information of at least 3 subjects with at least 2 weeks of daily dosing with rAvPAL-PEG. Initiation of dosing at higher or lower dose levels will be per the determination of the Sponsor's Medical Officer in consultation with the Investigator.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PKU with both of the following: current blood Phe concentration of ≥ 600 micromol/L at screening and average blood Phe concentration of ≥ 600 micromol/L over the past 3 years, using available data
* Evidence that the subject is a non-responder to Kuvan® treatment (ie, 4 weeks of treatment with 20 mg/kg/day of Kuvan, insufficient response per investigator determination, and treatment end date ≥ 14 days prior to Day 1 [ie, first dose]). Subjects who have had a previous response to Kuvan® treatment but are not currently taking Kuvan® because of noncompliance and have been off treatment for ≥ 4 months prior to screening are eligible for participation.
* Willing and able to provide written, signed informed consent, or, in the case of participants under the age of 18, provide written assent (if required) and written informed consent by a legally authorized representative, after the nature of the study has been explained, and prior to any research-related procedures.
* Willing and able to comply with all study procedures.
* Between the ages of 16 and 70 years, inclusive.
* Negative pregnancy test at screening and willing to have additional pregnancy tests performed during the study for females of childbearing potential only. Females considered not of childbearing potential are those who have been in menopause for at least 2 years or have had a tubal ligation at least 1 year prior to screening, or who have had a total hysterectomy.
* Willing to use an acceptable method of contraception while participating in the study (sexually active subjects only).
* Maintained a stable diet with no significant modifications during the 4 weeks preceding the administration of study drug.
* In generally good health as evidenced by physical examination, clinical laboratory evaluations (hematology, chemistry, and urinalysis), and ECG at screening.

Exclusion Criteria:

* Prior use of rAvPAL-PEG.
* Use of any investigational product or investigational medical device within 30 days prior to screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
* Use of any medication that is intended to treat PKU within 14 days prior to the administration of study drug.
* Use or planned use of any injectable drugs containing PEG (other than rAvPAL-PEG), including Depo-Provera, within 3 months prior to screening and during study participation.
* Known hypersensitivity to rAvPAL-PEG excipients.
* Breastfeeding at screening or planning to become pregnant (self or partner) or to breastfeed at any time during the study.
* Concurrent disease or condition that would interfere with study participation or safety (eg, history or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurological, oncologic, or psychiatric disease).
* Any condition that, in the view of the investigator, places the subject at high risk of poor treatment compliance or of not completing the study.
* Alanine aminotransferase (ALT) concentration > 2 times the upper limit of normal.
* Creatinine > 1.5 times the upper limit of normal.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ari Gershman, MD, Study Director — BioMarin Pharmaceutical
Locations (9):
- United States (9):
  - The Children's Hospital, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - Weisskopf Child Evaluation Center / University of Louisville, Louisville, Kentucky
  - University of Missouri, Columbia, Missouri
  - Washington University Center for Applied Research Sciences, St Louis, Missouri
  - Albany Medical Center, Albany, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Wisconsin-Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Burton BK, Longo N, Vockley J, Grange DK, Harding CO, Decker C, Li M, Lau K, Rosen O, Larimore K, Thomas J; PAL-002 and PAL-004 Investigators. Pegvaliase for the treatment of phenylketonuria: Results of the phase 2 dose-finding studies with long-term follow-up. Mol Genet Metab. 2020 Aug;130(4):239-246. doi: 10.1016/j.ymgme.2020.06.006. Epub 2020 Jun 16. PMID 32593547

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | rAvPAL-PEG
Started | 16
Completed | 15
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | rAvPAL-PEG
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.2 (8.27)
Age, Customized [Count of Participants; unit: Participants]
  < 18 years of age | 0
  > or = 18 years of age | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  Other | 0

OUTCOME MEASURES:

1. Primary Outcome: Blood Phenylalanine Concentration
Description: Plasma Phe
Time Frame: Baseline, Week 16
Population: The efficacy population will consist of all subjects who received any amount of study drug and have post-treatment blood Phe concentration measurements.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | rAvPAL-PEG
Number analyzed (Participants) | 16
umol/L
  Baseline | 1482.1 (363.46)
  Week 16 | 1566.0 (586.11)

2. Secondary Outcome: Study Drug Related Adverse Events
Description: Safety will be evaluated on the incidence of AEs and clinically significant changes in vital signs as well as clinical labs and ECG. Please refer to AE section below for comprehensive listing of all adverse events recorded during study.
Time Frame: Weekly
Population: The safety population will consist of all subjects who receive any amount of study drug throughout the study duration and have post-treatment safety information (laboratory values, vital signs, adverse events, 12-lead electrocardiogram, chest x-ray, antibodies, and physical examinations).
Measure: Count of Participants; unit: Participants
Groups:
- Total: The safety population will consist of all subjects who receive any amount of study drug throughout the study duration and have post-treatment safety information (laboratory values, vital signs, adverse events, 12-lead electrocardiogram, chest x-ray, antibodies, and physical examinations).
Arm/Group | Total
Number analyzed (Participants) | 16
Participants | 16

3. Secondary Outcome: Percentage of Participants With PAL IgG Antibody Percentage of Participants With Positive PAL IgG
Description: Antibody against phenylalanine ammonia lyase (PAL)
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Number; unit: Percentage
Groups:
- Total: rAvPAL-PEG in all doses.
Arm/Group | Total
Number analyzed (Participants) | 16
Percentage
  Baseline | 12.5
  Week 16 | 100.0

4. Secondary Outcome: Plasma Concentrations of rAvPAL-PEG (BMN 165)
Description: Measurements taken pre-dose
Time Frame: Baseline, Week 8, Week 13
Population: The PK population will consist of all subjects who received any amount of study drug and have post-treatment plasma BMN 165 concentration measurements.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | rAvPAL-PEG
Number analyzed (Participants) | 16
ng/mL
  Baseline-Day 1, 1 Hour Predose | 0.000 (0.0000)
  Week 8-Day 52, 1 Hour Predose | 2425.608 (8532.2431)
  Week 13-Day 89, Predose | 1116.364 (2013.9676)

5. Secondary Outcome: Percentage of Participants With PEG-IgG Antibody Positivity
Description: Antibodies against polyethylene glycol (PEG) of the IgG isotype
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Number; unit: Percentage
Arm/Group | Total
Number analyzed (Participants) | 16
Percentage
  Baseline | 25.0
  Week 16 | 75.0

6. Secondary Outcome: Percentage of Participants With PAL-IgM Antibody Positivity
Description: Antibodies against phenylalanine ammonia lyase (PAL) of the IgM isotype
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Number; unit: Percentage
Arm/Group | Total
Number analyzed (Participants) | 16
Percentage
  Baseline | 12.5
  Week 16 | 75.0

7. Secondary Outcome: Percentage of Participants With PEG-IgM Antibody Positivity
Description: Antibodies against polyethylene glycol (PEG) of the IgM isotype
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Number; unit: Percentage
Arm/Group | Total
Number analyzed (Participants) | 16
Percentage
  Baseline | 31.3
  Week 16 | 50.0

8. Secondary Outcome: Percentage of Participants With Neutralizing Antibody Positivity
Description: Antibody positivity over time
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Number; unit: Percentage
Arm/Group | Total
Number analyzed (Participants) | 16
Percentage
  Baseline | 0.0
  Week 16: number analyzed (Participants) | 4
  Week 16 | 0.0

9. Secondary Outcome: Percentage of Participants With PAL-IgE Antibody Positivity
Description: Antibodies against phenylalanine ammonia lyase (PAL) of the IgE isotype
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Number; unit: Percentage
Arm/Group | Total
Number analyzed (Participants) | 16
Percentage
  Baseline | 0.0
  Week 16 | 0.0

10. Secondary Outcome: Percentage of Participants With PAL-PEG-IgE Antibody Positivity
Description: Antibodies against phenylalanine ammonia lyase (PAL)-polyethylene glycol (PEG) of the IgE isotype
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Number; unit: Percentage
Arm/Group | Total
Number analyzed (Participants) | 16
Percentage
  Baseline | 0.0
  Week 16 | 0.0

ADVERSE EVENTS:
Time Frame: Week 0- Week 16
Arm/Group | rAvPAL-PEG
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 1/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rAvPAL-PEG (N=16)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rAvPAL-PEG (N=16)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (2)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Ear pruritus (Ear and labyrinth disorders) | 1 (1)
Motion sickness (Ear and labyrinth disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Ocular hyperaemia (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (9)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 4 (5)
Flatulence (Gastrointestinal disorders) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (5)
Toothache (Gastrointestinal disorders) | 1 (1)
Chest discomfort (General disorders) | 3 (3)
Chills (General disorders) | 3 (4)
Fatigue (General disorders) | 2 (2)
Hangover (General disorders) | 1 (1)
Infusion site erythema (General disorders) | 2 (8)
Injection site bruising (General disorders) | 6 (11)
Injection site erythema (General disorders) | 8 (18)
Injection site induration (General disorders) | 1 (2)
Injection site nodule (General disorders) | 1 (1)
Injection site oedema (General disorders) | 1 (1)
Injection site pain (General disorders) | 7 (9)
Injection site pruritus (General disorders) | 1 (1)
Injection site rash (General disorders) | 4 (8)
Injection site reaction (General disorders) | 8 (32)
Injection site swelling (General disorders) | 1 (1)
Injection site urticaria (General disorders) | 4 (10)
Injection site warmth (General disorders) | 2 (3)
Instillation site pruritus (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (6)
Oedema peripheral (General disorders) | 2 (2)
Pain (General disorders) | 1 (2)
Pyrexia (General disorders) | 5 (6)
Swelling (General disorders) | 1 (1)
Vessel puncture site bruise (General disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2)
Pharyngitis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
C-reactive protein increased (Investigations) | 3 (3)
Complement factor C3 decreased (Investigations) | 3 (3)
Complement factor C4 decreased (Investigations) | 2 (2)
Complement factor decreased (Investigations) | 1 (1)
Complement factor increased (Investigations) | 1 (1)
Electrocardiogram ST segment depression (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (36)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 2 (3)
Joint swelling (Musculoskeletal and connective tissue disorders) | 4 (5)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (6)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (5)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Burning sensation (Nervous system disorders) | 1 (1)
Clonus (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 9 (14)
Dizziness postural (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 10 (34)
Hyperreflexia (Nervous system disorders) | 2 (2)
Hypersomnia (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 3 (5)
Paraesthesia (Nervous system disorders) | 2 (3)
Sciatica (Nervous system disorders) | 1 (1)
Sinus headache (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 4 (5)
Anxiety (Psychiatric disorders) | 1 (1)
Nervousness (Psychiatric disorders) | 1 (1)
Uterine spasm (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hypopnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 2 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (9)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Rash erythematous (Skin and subcutaneous tissue disorders) | 3 (3)
Rash generalised (Skin and subcutaneous tissue disorders) | 6 (7)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (3)
Endodontic procedure (Surgical and medical procedures) | 1 (2)
Flushing (Vascular disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days